CLINICAL TRIAL: NCT04756895
Title: Vancomycin Dose Adjustments Comparing Trough Levels to The AUC0-24h/MIC Method Using a Bayesian Approach in a Hospitalized Adult Population: A Pilot Study
Brief Title: Vancomycin Dose Adjustments Comparing Trough Levels to The AUC/MIC Method Using a Bayesian Approach in a Hospitalized Adult Population
Acronym: VancoDATABayes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CR-CSSS Champlain-Charles-Le Moyne (Other)
Responsible Party: Principal Investigator, Benoit Crevier, Principal Investigator, CR-CSSS Champlain-Charles-Le Moyne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-600
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Vancomycin; Adult; Area Under Curve
Keywords: Bayesian approach; Dose adjustments; trough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bayesian method (Experimental): Pharmacists will perform vancomycin dose adjustments according to AUC0-24h/MIC using the Bayesian method with a web application
  Interventions: Other: Vancomycin dose adjustment using the Bayesian method
- Standard method (Active Comparator): Pharmacists will perform vancomycin dose adjustments according to trough levels of vancomycin.
  Interventions: Other: Vancomycin dose adjustment using the trough level method

INTERVENTIONS:
Other: Vancomycin dose adjustment using the Bayesian method — This intervention is the experimental method. The AUC/MIC target is 400-600 mg*hour/L.
  Arms: Bayesian method
Other: Vancomycin dose adjustment using the trough level method — This intervention is the standard method. Previous clinical guidelines recommended this method. The trough target is 10-15 mg/L for non-severe infections and 15-20 mg/L for severe infections.
  Arms: Standard method

SUMMARY:
This pilot study is a prospective, randomized, controlled, open-label trial to assess the feasibility of a randomized controlled trial of sufficient quality that would assess the efficacy and safety of vancomycin adjustments according to Area under the curve/Minimal inhibitory concentration (AUC0-24h/MIC) calculated by the Bayesian approach rather than by a trough dosage. Randomization will be stratified according to infection severity. Approximately 60 subjects meeting all inclusion and no exclusion criteria will be randomized to have pharmacists perform vancomycin dose adjustments with AUC0-24h / MIC calculated by the Bayesian approach versus the trough dosage approach.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Hospitalized patients
* Suspected or confirmed infection;
* Anticipated IV vancomycin treatment for 24 hours or more.

Exclusion Criteria:

* Patients with renal replacement therapy (peritoneal dialysis, continuous renal replacement therapy or hemodialysis);
* Treatment of vancomycin in continuous infusion;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Validation of The Research Protocol | Through study completion, an average of 2 weeks
  Evaluation of adhesion rate to the sampling protocol of 80% or more and adhesion rate to software recommendations of 90% or more
Evaluation of Recruitment | Baseline
  Evaluation of consent rate of 30% or more and the number of patients recruited per month of 10 or more

SECONDARY OUTCOMES:
The proportion of patients who reach a therapeutic level in the first 48 hours | At 48 hours after the first dose of vancomycin
  Percentage of patients who reach a therapeutic level in the first 48 hours
Time to reach the vancomycin target | During the vancomycin treatment
  Number of hours necessary to reach the vancomycin target. Number of hours will be classified in the following categories: 24-48 hours, 49-96 hours, 97 hours and above.
The number of adjustments required to reach the vancomycin target | During the vancomycin treatment
  Number of dose adjustments required to reach the vancomycin target
The number of vancomycin dosage level monitoring to reach the vancomycin target | During the vancomycin treatment
  The number of vancomycin dosage level monitoring to reach the vancomycin target
The proportion of vancomycin dosage level monitoring in the vancomycin target | During the vancomycin treatment
  Percentage of vancomycin dosage level monitoring in the vancomycin target
The difference between the AUC calculated by the Bayesian method and the trapezoid method | During the vancomycin treatment
  Difference in percentage of the vancomycin AUC calculated by the Bayesian method and the trapezoid method
The difference between the initial prescribed dose and the dose suggested by the Bayesian software. | Baseline
  Difference in percentage of the initial prescribed dose and the dose suggested by the Bayesian software.
Proportion of acute kidney injury | During the vancomycin treatment
  Percentage of acute kidney injury.
Average daily dose of vancomycin | Through study completion, an average of 2 weeks
  Average of the daily dose of vancomycin calculated in mg per kg of total body weight
Operational Impact | Immediately after the intervention
  Evaluation of the impact on pharmacist's time required for monitoring vancomycin

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Crevier, PharmD, MSc, Principal Investigator — Charles-Le Moyne Hospital
Locations (1):
- Charles-Le Moyne Hospital, Greenfield Park, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No